CLINICAL TRIAL: NCT03935347
Title: Phase 2 Study of Autologous Tumor Infiltrating Lymphocytes (LN-145) With Pembrolizumab, in Subjects Who Have Failed Cisplatin-Based Chemotherapy With Locally Advanced (Unresectable) or Metastatic Transitional Cell Cancer (TCC) of the Urothelium
Brief Title: Adoptive Cell Therapy With (LN-145) in Combination With Pembrolizumab in Treating Patients With Unresectable or Metastatic Transitional Cell Cancer Who Have Failed Cisplatin-Based Chemotherapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 77218; P30CA16056OD (Other Grant/Funding Number: NCI); P30CA016056 (NIH)
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Metastatic Bladder Urothelial Carcinoma; Metastatic Renal Pelvis Urothelial Carcinoma; Metastatic Ureter Urothelial Carcinoma; Metastatic Urethral Urothelial Carcinoma; Unresectable Renal Pelvis Urothelial Carcinoma; Unresectable Ureter Urothelial Carcinoma
MeSH Terms: interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; pembrolizumab; Immunoglobulin G; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cyclophosphamide, fludarabine, pembrolizumab) (Experimental): Patients receive cyclophosphamide IV over 2 hours on days -8 and -7, fludarabine IV over 30 minutes on days -6 to -2, and pembrolizumab IV over 30 minutes on day -1. At least 24 hours later, patients receive autologous tumor infiltrating lymphocytes LN-145 IV on day 0, and receive aldesleukin IV over 30 minutes for up to 6 doses on days 1-4. Patients then continue receiving pembrolizumab IV over 30 minutes beginning on day 21. Cycles of pembrolizumab repeat every 21 days for 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Fludarabine Phosphate; Biological: Pembrolizumab; Biological: Autologous Tumor Infiltrating Lymphocytes LN-145; Biological: Aldesleukin

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: 1-bis(2-chloroethyl)-amino-1-oxo-2-aza-5-oxaphosphoridin monohydrate; 2-[bi(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate; Cyclostine; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: 118218; 2-Fluoro-9-beta-arabinofuranosyladenine; 2-Fluorovidarabine, 21679-14-1; 9-Beta-D-arabinofuranosyl-2-fluoro-9H-purin-6-amine; 9-Beta-D-arabinofuranosyl-2-fluoroadenine; Fluradosa
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 312887; 328002; 75607-67-9; 9H-Purin-6-amine; 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl; Fludarabine-5'-Monophosphate; SH T 586
Biological: Pembrolizumab — Given IV
  Other Names: 1374853-91-4; Immunoglobulin G4; Anti-(Human Programmed Cell Death 1)
Biological: Autologous Tumor Infiltrating Lymphocytes LN-145 — Given IV
  Other Names: Autologous TILs LN-145; LN-145; LN145
Biological: Aldesleukin — Given IV
  Other Names: 110942-02-4; 125-L-Serine-2-133-interleukin 2; Recombinant Human Interleukin-2

SUMMARY:
This phase II trial studies how well autologous tumor infiltrating lymphocytes (LN-145) and pembrolizumab work in treating patients with transitional cell cancer that cannot be removed by surgery or has spread to other places in the body and have failed cisplatin-based chemotherapy. LN-145 is made up of specialized immune cells called lymphocytes or T cells that are taken from a patient's tumor, grown in a manufacturing facility and infused back into the preconditioned patient to attack the tumor. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving LN-145 may help control transitional cell bladder cancer when given together with pembrolizumab

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of autologous tumor infiltrating lymphocytes LN-145 (LN-145) in combination with pembrolizumab in subjects with advanced transitional cell bladder cancer (TCC) using the objective response rate (ORR) and the duration of response (DoR), using the Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST version [v] 1.1).

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of LN-145 in combination with pembrolizumab in subjects with TCC based on the progression-free survival (PFS) and overall survival (OS).

II. To evaluate the safety of LN-145 in combination with pembrolizumab in subjects with TCC based on the adverse event (AE) profile per Common Terminology Criteria for Adverse Events, version 5.0 (CTCAE v5.0).

ELIGIBILITY:
Inclusion Criteria:

* The subject must understand the requirements of the study and voluntarily sign the informed consent form (ICF)
* All subjects must have a histologically confirmed unresectable TCC (including renal pelvis, ureters, urinary bladder, and urethra)
* Failed one and only one line of cisplatin-based chemotherapy per FDA guidelines.
* Subjects must have an area of tumor amenable to excisional biopsy for the generation of TIL separate from, and in addition to , a target lesion to be used for response assessment.Have at least one resectable lesion to generate TILs
* At least one measurable target lesion as defined by RECIST version 1.1
* An Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* Estimated life expectancy of >= 6 months
* Adequate bone marrow function
* Adequate organ function
* Subjects must be seronegative for the human immunodeficiency virus (HIV)
* Recovered from all prior anticancer therapy-related AEs to grade 1 or less
* Negative serum pregnancy test (female subjects of childbearing potential)
* Subjects of childbearing potential must be willing to practice an approved method of birth control starting at the time of informed consent and for 12 months after the completion of the study treatment regimen
* Must be able and willing to comply with the study visit schedule and protocol requirements including long-term follow-up

Exclusion Criteria:

* Have had another primary malignancy within the previous 3 years (with the exception of carcinoma in situ of the breast, cervix, or localized prostate cancer and non-melanoma skin cancer that has been adequately treated)
* Have received prior cell transfer therapy that included a nonmyeloablative or myeloablative chemotherapy regimen
* Prior treatment with anti-PD-1, or anti-PD-L1 therapeutic antibody, or pathway-targeting agents
* Chemotherapy or radiotherapy with projected completion within 4 weeks of initiating study treatment
* Bisphosphonate therapy for symptomatic hypercalcemia
* Have had treatment with systemic immunostimulatory agents (including, but not limited to, interferon [IFN]-alpha or interleukin [IL]-2) within 6 weeks before initiation of study treatment
* Active or prior documented autoimmune or inflammatory disorders
* Subjects who have any form of human immondeficiency virus (HIV)infection
* Have severe infections within 4 weeks before initiation of study treatment
* Have received a live or attenuated vaccine within 28 days of the non-myeloablative lymphodepletion (NMA-LD regimen)
* Subjects with a history of hypersensitivity reaction(s) to any component of the LN-145 therapy and/or the other study drugs

  * Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) >= 450 msec for males (and >= 470 msec for females) calculated from 3 electrocardiograms (ECGs) (within a 30-minute timeframe) or history of familiar long-QT syndrome
* Subjects who have a left ventricular ejection fraction (LVEF) < 45% or who are New York Heart Association functional classification class II or higher
* Serious illnesses or medical conditions, which would pose increased risk for study participation and/or compliance with the protocol
* Known clinically significant liver disease
* Have obstructive or restrictive pulmonary disease and have a documented FEV1 (forced expiratory volume in 1 second) of =< 60%
* Subjects with known primary central nervous system (CNS) malignancy or symptomatic CNS metastases
* Subjects who are pregnant or breastfeeding
* Active infection including tuberculosis (TB), hepatitis B, hepatitis C, or human immunodeficiency virus
* Treatment with any other investigational agent within 4 weeks before initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 3 years
  The proportion of subjects who achieve either a confirmed partial response (PR) or complete response (CR) as best response as assessed per Response Evaluation Criteria in Solid Tumors 1.1. Will be evaluated per each disease assessment and calculated with the corresponding 95% two-sided confidence interval

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | From the first dose of cyclophosphamide up to 30 days from the last dose of IL-
  Will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 5 by grade of severity and relationship to the study treatment.
Duration of response | Up to 3 years
  Will be assessed by Kaplan-Meier methods
Disease Control Rate | Up to 3 years
  Derived as the sum of the number of subjects who achieved confirmed PR/CR or sustained stable disease (at least 6 weeks) divided by the number of subjects in the all-treated population x 100%. Will be assessed by Kaplan-Meier methods
Progression-free survival | Up to 3 years
  Will be assessed by Kaplan-Meier methods
Overall Survival | Up to 3 years
  From time of lymphodepletion to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Gurkamal Chatta, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No